CLINICAL TRIAL: NCT01885546
Title: Accuracy Study for the Evaluation of Obtaining an Enhanced Meter Feature Using an AgaMatrix BGMS
Brief Title: Accuracy Study for Enhanced Meter Feature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AgaMatrix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AGAFPGM02
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; glucose; glucometer
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enhanced meter feature usability (Other): Home diabetes monitoring by patient using provided blood glucose monitoring system.
  Interventions: Device: AgaMatrix Blood Glucose Monitor

INTERVENTIONS:
Device: AgaMatrix Blood Glucose Monitor

SUMMARY:
This enhanced meter feature raises awareness among patients by providing additional information regarding their glycemic control between Healthcare Professional visits. This information may facilitate increased dialogue between patient and Healthcare Professionals and can remind patients of the importance of glycemic control.

This study will evaluate a user's ability to obtain the enhanced meter feature.

ELIGIBILITY:
Inclusion Criteria:

* Type I or type II diabetes inclusive of the following populations:

  1. Mixed insulin therapies
  2. Basal insulin therapies
  3. Continuous subcutaneous insulin infusion therapies
  4. Multiple daily injection therapies
  5. Non-insulin diabetic treatments (oral and injectable)
  6. Life style (exercise and diet) diabetes management
  7. New diagnosis of diabetes
* Non diabetics
* Able to speak and read English proficiently
* Subjects must be willing to:

  1. once a month, perform a 7 point blood glucose profile over the course of one day
  2. perform fasting blood glucose tests every day
  3. complete baseline and follow-up questionnaires
  4. consent to baseline HbA1c assays

Exclusion Criteria:

* Pregnant
* Hct <20 or >60
* Work for BGM competitor company (including, but not limited to Lifescan, Roche, Abbott)
* Homeless
* Incarcerated
* Mentally ill
* Employees or students of the Research Site, including the Principal Investigator, directly involved in the conduct of the protocol.
* Has any condition that the Principal Investigator believes may interfere in the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
User's ability to obtain the enhanced meter feature | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- MassResearch, LLC, Waltham, Massachusetts, United States

REFERENCES:
- [Derived] Sieber J, Flacke F, Dumais B, Peters CC, Mallery EB, Taylor L. Evaluation of a Methodology for Estimating HbA1c Value by a New Glucose Meter. J Diabetes Sci Technol. 2015 May 22;10(1):67-71. doi: 10.1177/1932296815587323. PMID 26002835